CLINICAL TRIAL: NCT04623060
Title: Feasibility of Low-Volume Interval Training and Resistance Exercise on Walking Performance, Aerobic Fitness, Muscle Strength and Quality Of Life in Individual With Stroke
Brief Title: Low-Volume Interval Training and Resistance Exercise in Individual With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Mohd Haidzir Abd Manaf, Associate Professor, Universiti Teknologi Mara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/401/19
Record Dates: First submitted 2020-10-20; First posted 2020-11-10 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Stroke
Keywords: Low-Volume Interval Training; Resistance Training
MeSH Terms: conditions — Stroke | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 3 sessions/week for 6 weeks
  Interventions: Other: Combination of Low-volume interval treadmill training and Resistance Training

INTERVENTIONS:
Other: Combination of Low-volume interval treadmill training and Resistance Training — Low-volume interval training (LV-ITT) protocols included a 5 min warm-up (30%-50%VO2peak) up to 20min of LV-ITT and a 5 min cooling down (30%-50% VO2peak). The LV-ITT will repeat 60s bursts of fast treadmill walking at maximum tolerate speed (0% incline), alternate with pre-specified recovery periods about 4 minutes according to protocol. Each time the participants completed a burst successfully, treadmill speed will be increased by 0.1 mph for the next burst. The recovery periods will be 4 minutes. The intervention will be conducted for about 30 minutes.
  Resistance training will be conducted by using a horizontal leg press machine. They are encouraged to focus on an explosive concentric movement and a controlled eccentric movement such that the time on each phase was in the ratio 1:2.

SUMMARY:
To examine the feasibility of Low-Volume Interval Training (LV-ITT) and Resistance Exercise (RE) on walking performance (walking endurance, gait speed, functional balance), lower limb muscle strength and quality of life among individuals with post-stroke.

DETAILED DESCRIPTION:
Prescribing aerobic and resistance training in concurrence is proposed as an optimum strategy to target cardiovascular as well as musculoskeletal functions in individuals with post-stroke. Lower limb's resistance training alone in chronic stroke produces a large effect on muscle strength. However, it has shown uncertainty results on walking performance. Therefore, it is suggested that to prescribe mix training (treadmill training and strength training) in order to improve muscle strength, gait performance and quality of life in stroke survivors. Previous studies have shown the effect of mixed training on walking performance and endurance in other populations such as multiple sclerosis and coronary artery disease. However, there is a lack of study that conducted mixed training among chronic post-stroke. Therefore, the feasibility study on the effectiveness of combining LV-ITT and RE in post-stroke should be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 45-65 years' old
* At least 3-months post-stroke
* Gait speed ≤1.0 m·s -¹ measured by the 10 m walk test.
* Able to walk 10 m overground with assistive devices as needed and no physical assistance.
* Able to walk for 3 min on the treadmill at ≥0.17 m·s -¹ (0.4 mph) with no aerobic exercise contraindications.
* Modified Rankin Score (mRS) of <4 at the screening
* American Heart Association class B (2), allowing for aerobic capacity <6 metabolic equivalent (MET)

Exclusion Criteria:

* Significant resting ECG abnormalities
* Hospitalization for cardiac or pulmonary disease within 3 months
* Using Pacemaker
* Aphasia
* Significant musculotendinous or bony restrictions of the affected limb, or any serious chronic disease independently causing disability or profound atrophy of the affected limb that will comprise further indications to participation significant.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Six Minute Walk Test | 0, 6 weeks
  This test measures the distance that an individual can quickly walk in a period of 6 minutes on a flat surface. Participants will complete one trial with the gait aide prescribed to them. The distance will be recorded. Participants can stop and rest or discontinue to the test at any time.

SECONDARY OUTCOMES:
Change in 10-meter walk test | 0, 6 weeks
  This assessment will include four 10-meter walking tasks at maximal comfortable speed.
Change in Lower Limb Muscle Strength | 0, 6 weeks
  Handheld dynamometer for knee extensor
Change in Timed Up and Go test | 0, 6 weeks
  Functional Balance
Stroke Impact Scale (SIS) | 0,week 6
  Quality of Life
Adherence | 0 to 6 weeks
  Attendance and completion of home-based sessions measured via exercise diary
Adverse Events | 0 to 6 weeks
  Any adverse event or near miss is required to be reported as standard of care at Selayang Hospital
Patient satisfaction | 6 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Haidzir Abd Manaf, PhD, Principal Investigator — Universiti Teknologi Mara
Locations (1):
- Hospital Selayang, Batu Caves, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No